CLINICAL TRIAL: NCT05754398
Title: Measuring the Effects of a Nurse-led Intervention on Frailty Status of Older Persons Living in the Community in Ethiopia: A Protocol for a Quasi-experimental Study
Brief Title: A Nurse-led Intervention on Frailty Status of Ethiopian Older Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wollongong (Other)
Responsible Party: Principal Investigator, Ayele Semachew Kasa, Principal Investigator, University of Wollongong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022/212
Record Dates: First submitted 2023-02-10; First posted 2023-03-03 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Frailty
Keywords: Nurse-led; Intervention; Frailty; Elderly; Ethiopia
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: A single-group pre-, post-, and follow-up single-group quasi-experimental study design will be adopted to examine the effect of a nurse-led intervention on frailty among older persons living in Bahir Dar City, Ethiopia.
Masking Description: The data will be collected through a face-to-face administered structured survey questionnaire, and anthropometrical physical measurements. To reduce assessor bias, CHWs will not be involved in the data collection process. Hence, two professional nurses from Bahir Dar city will be recruited for data collection. The data collectors will not be involved in providing the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group will receive the nurse-led intervention (Other): A single group of community-dwelling older persons will receive a nurse-led intervention after an initial screening and eligibility checks.
  Interventions: Behavioral: six independent and interconnected educational training sessions

INTERVENTIONS:
Behavioral: six independent and interconnected educational training sessions — Each of the six components will be offered each month for six consecutive months. Each session will last approximately 30 to 40 minutes.
  All the six sessions will be delivered through a face-to-face approach.

SUMMARY:
The goals of this study are to design, implement, and evaluate the effects of a nurse-led intervention on the frailty and quality of life of older persons living in the community in Ethiopia. The main hypothesis aims to test the following:

1. Effects of a nurse-led intervention on frailty, including physical, social, and psychological domains of older persons living in the community in Bahir Dar, Ethiopia.
2. Effects of a nurse-led intervention improve the quality of life among the older persons living in the community of Bahir Dar, Ethiopia.

The nurse-led intervention consists of six independent interconnected education sessions focused on specific topic areas consisting of ageing and age-related changes, healthy nutrition, physical activity, mental health, social interaction, and support, and lastly an overall discussion on the intervention. The intervention is delivered one-on-one and face-to-face to the family homes of older people living in the community by specialist nurses who are community health workers (CHWs). Each CHW will be provided with a notebook to record the progress of each participant undertaking the program and any questions that need to be followed up at a subsequent session.

DETAILED DESCRIPTION:
The intervention consists of six independent interconnected education sessions focused on specific topic areas: ageing and age-related changes, healthy nutrition, physical activity, mental health, social interaction and support, and overall discussion.

A specialist community nurses will deliver the intervention. In each session, the nurse will describe the education, including its learning objectives, ask leading questions of the start of each session, and at the end of each session the participants will be provided with a simple take-home message on the specific topic discussed. The participants will have the opportunity to reflect on ideas, ask questions and discuss with the nurses delivering the intervention.

Session 1: Ageing and age-related changes

* Age and age-related changes,
* Sensory and perceptual changes on older persons
* Other changes that may happen in later life Session 2: Healthy nutrition
* Healthy diet for older persons
* Factors that cause nutritional problems in older persons
* Nutritional needs of older persons Session 3: Physical activity
* The need for physical activity for an older person
* The types of exercises that older people need to do
* How older people initiate exercise in a safe way Session 4: Mental health
* Ageing and mental health
* Factors for mental health problems in older persons
* Strategies to improve mental well-being in older persons Session 5: Social interaction and support
* The need for social participation and support
* The Risks of Senior Isolation Session 6: Overall discussion session
* This is the last session focused on an overall discussion and reflection with each study participant about the previous sessions.
* Discussion will also be made on how the study participants will sustain and implement the intervention in their day-to-day activities in their future life. To measure adherence to the program the CHWs will maintain an attendance record. At the beginning of each session the CHWs will record attendance of the participants by checking off the name of a participant against each session in their notebook. Acceptability of the program from the perspectives of the CHWs will be recorded in two ways: (1) field notes written by the CHWs in the notebooks they used to while delivering the program and (2) at the end of the intervention. The informal discussions with the CHWs will also be used to generate feedback about the training handbook.

The six sessions will be delivered over six consecutive months with each monthly session focusing consecutively on each the specific intervention topics. Each session will last approximately 30 to 40 minutes.

The intervention will be delivered by two community health workers (CHWs) under the supervision and support of the nursing Ph.D. candidate leading this study.

All six sessions will be delivered one-on-one and face-to-face in the home of the participants. During the six months when the intervention is delivered, there will be a fortnightly 5 to 10-minute follow-up phone call with participants to receive feedback about the education sessions and provide opportunistic counseling on the specific topics.

At the end of each education session, participants will be provided with a simple but relevant take-home message about the specific session topic. At the end of each session the CHW will be required to reflect on how each participant undertakes their take-home message and commence the subsequent education session from the reflection. If a participant asks questions beyond the scope of the intervention material, depending on the nature of the question, they will be advised to meet with a medical expert at a nearby healthcare facility.

To reduce loss to follow-up (LTFU) and increase adherence rates to intervention, participants will be encouraged and reminded by phone to attend upcoming sessions. The study construct of the Nurse-led Intervention (NLI) is indicated below.

CHWs are registered nurses employed by the local government and work closely with the local community home-to-home and at health posts. CHWs know the culture, lifestyle, and social norms of the community and provide culturally appropriate health education and information, help community members access the care they need, counsel and guide on health-promoting behaviours, and for the health needs of individuals and communities.

ELIGIBILITY:
Inclusion Criteria:

* In Ethiopia, the cut points of old age started at 60 years.
* Older persons aged 60 years or above.
* Older persons whose frailty score is ≥ 5 as measured by the Tilburg Frailty Indicator (TFI).
* Older persons residing in Bahir Dar, Ethiopia.

Exclusion Criteria:

Older persons who:

* are unable to communicate.
* have a cognitive impairment.
* are bed-redden.
* are not living at home.
* have been hospitalised with a known psychiatric problem within the past six months, and
* will not remain in the selected area during the study period.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Change in frailty status of community-dwelling older persons. | Change in frailty will be measured at baseline (before intervention) (T0), immediately after the intervention (T1) and at twelfth week of the intervention
  Changes in frailty will be measured using the Tilburg Frailty Indicator (TFI). The TFI comprises 15 self-reported questions, divided into three distinct domains. The physical, psychological, and social domains are the three distinct domains that constitute the TFI. The physical domain consists of eight questions related to different physical health of older persons. The psychological domain contains four items related to the psychological health of older persons. The last domain, the social domain has three questions related to social relations. Eleven items of the TFI have two response categories as "yes" or "no" options, while three items from the psychological domain and one item from the social domain have three response categories as "yes", "no," or "sometimes". The instrument's total score ranges from 0 to 15: the higher the score, the higher one's frailty. Frailty is diagnosed when the total TFI score is ≥5.

SECONDARY OUTCOMES:
Change in the activity of daily living of community-dwelling older persons. | Changes in activity of daily living will be measured at baseline (before intervention) (T0), immediately after the intervention (T1) and at twelfth week of the intervention
  The activity of daily living will be measured using the Katz Index of Independence in Activities of Daily Living. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. The responses are scored as a 'Yes' or 'No' for independence in each of the six functions. The minimum and maximum scores are 0 (zero) and 6 (six) respectively. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Change in the nutritional status of community-dwelling older persons. | Change in nutritional status will be measured at baseline (before intervention) (T0), immediately after the intervention (T1) and at twelfth week of the intervention
  Changes in nutritional status will be measured using the Mini-Nutritional Assessment (MNA) tool. The MNA score ranges from 0 to 30. A higher score indicates a better nutritional status. Moreover, based on the MNA score, the nutritional status of older persons will be classified as:
  Malnourished (MNA Score <17), At risk of malnutrition (MNA Score 17 to 23.5) or Normal nutritional status (MNA Score 24 to 30).
Change in the level of depression | Changes in depression status will be measured at baseline (before intervention) (T0), immediately after the intervention (T1) and at twelfth week of the intervention
  The Geriatric Depression rating Scale-15 (GDS-15) will be used to measure the changes in depression. The values range from 0 to 15: the higher the score, the higher one's depression. Depression is considered using a cutoff point greater than or equal to five. The outcome will be coded depending on the cutoff point 0 to 4 as normal, 5 to 8 as mild depression, 9 to 11 as moderate depression, and 12 to 15 as severe depression
Change in quality of life | Changes in quality of life will be measuredat baseline (before intervention) (T0), immediately after the intervention (T1) and at twelfth week of the intervention
  World Health Organization's Quality of Life Questionnaire (WHOQOL-BREF) will be used to measure the changes in quality of life of older persons. WHOQOL-BREF is a self-report questionnaire or interviewer-administered which contains 26 questions categorized into four domains that are scored on a 5-point Likert scale. The four domains are physical health (7 items), psychological health (6 items), social relationships (3 items), and environment (8 items). Values will be transformed into scores ranging from 0 to 100 according to the WHO guidelines. The higher the score the higher the quality of life. Two (question number 1 and 2) items measure the overall QOL and general health.
Change in height | Changes in height will be measured at baseline (before intervention) (T0), immediately after the intervention (T1) and at twelfth week of the intervention
  Change in height measurements will be taken without heavy outdoor clothing. Height will be measured using standard and caliber anthropometric rods in centimeters. In combination with the weight (in kg) of the study participant, the measured height then will be used to determine the Body Mass Index (BMI) of the study participant.
Change in weight | Changes in weight will be measured at baseline (before intervention) (T0), immediately after the intervention (T1) and at twelfth week of the intervention
  Changes in weight will be measured on a pre-standardized body weighing scale in kilograms. In combination with the height (in m2) of the study participant, the measured weight then will be used to determine the Body Mass Index of the study participant.
Change in Calf Circumference (CC) | Changes in calf circumference will be measured at baseline (before intervention) (T0), immediately after the intervention (T1) and at twelfth week of the intervention
  Calf Circumference (CC) will be measured using a tape meter in millimeters. The study participant will sit on a chair and hold his/her bare foot down, holding the leg folded to 90 degrees. The circumference of the calf at its widest point will be measured, laying the tape on the skin without tightening. The measurement will be taken at more than one point to ensure the measurement is taken at the widest part. An increased CC is associated with good nutrition status in older persons as measured in MNA.
Change in Body Mass Index (BMI) | Changes in Body Mass Index (BMI) will be measured at baseline (before intervention) (T0), immediately after the intervention (T1) and at twelfth week of the intervention
  Height & weight measures will be aggregated to report Body Mass Index (BMI) as Weight measured in kilograms divided by height in meter square i.e [ Weight (kg)/Height (m2)]. An increased BMI is associated with increased nutrition status in older persons.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Traynor, Professor, Study Director — University of Wollongong; Peta Drury, PhD, Study Chair — University of Wollongong; Shu-Chun Lee, PhD, Study Chair — Taipei Medical University; Hui-Chen (Rita) Chang, PhD, Study Chair — University of Wollongong
Locations (1):
- Bahir Dar University, Bahir Dar, Amhara, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The time frame will start from the time when summary data are published or start 6 months after publication.
Access Criteria: IPD and additional supporting data information will be shared with scientific communities, readers, and other interested bodies through open-access journals.

REFERENCES:
- [Derived] Kasa AS, Traynor V, Drury P. Measuring the effects of nurse-led frailty intervention on community-dwelling older people in Ethiopia: a quasi-experimental study. BMC Geriatr. 2024 Apr 30;24(1):384. doi: 10.1186/s12877-024-04909-2. PMID 38689218
- [Derived] Kasa AS, Drury P, Chang HR, Lee SC, Traynor V. Measuring the effects of a nurse-led intervention on frailty status of older people living in the community in Ethiopia: A protocol for a quasi-experimental study. PLoS One. 2024 Jan 19;19(1):e0296166. doi: 10.1371/journal.pone.0296166. eCollection 2024. PMID 38241265